CLINICAL TRIAL: NCT00251563
Title: Epidemiologic, Laboratory, and Clinical Characterization of Individuals With Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Other Study IDs: ICP036
Record Dates: First submitted 2005-11-09; First posted 2005-11-10 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2005-11

CONDITIONS: Cancer
Keywords: Cancer,Risk factors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Environmental and genetic factors may play a role in the progression of cancer. The goal of this project is to establish a series of cross-sectional / case-control studies to evaluate risk factors of cancer in China.

DETAILED DESCRIPTION:
This study is designed to investigate the epidemiologic, genetic, laboratory and clinical characterization of individuals with cancer (gastric, colorectal, esophageal, liver, prostate, lung, breast and endometrial cancer, etc.). We will accrue approximately 1600 patients as experimental group. The control group consists of subjects who will be confirmed without cancer. We will explore the environmental (including family history, life style, diet, physical activity, neuropsychological functioning，plasma levels of oxidative stress factors, angiogenic factors, and tumor markers, etc.) and genetic (including oxidative stress factors and angiogenic factors, etc.) risk factors. We will study the association between various environmental risk factors with the clinical characterization and correlation between the genetic polymorphisms and the presence of various cancer.

ELIGIBILITY:
Inclusion Criteria:

* This is a study only of Chinese. Subjects will be allowed to participate if they self-identify as Chinese. The age range of the participants will be between 18 and 89 years. Individuals with cancer (gastric, colorectal, esophageal, liver, prostate, lung, breast and endometrial cancer, etc.) will be allowed to participate. To participate in the study as the control, subjects should be confirmed without cancer.

Exclusion Criteria:

-

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Bin Wang, Ph.D, Principal Investigator — Department of Pharmacology, Institute of Clinical Pharmacology, Nanjing Medical University
Locations (1):
- Department of Pharmacology, Institute of Clinical Pharmacology, Nanjing Medical University, Nanjing, Jiangsu, China